CLINICAL TRIAL: NCT06344793
Title: A Multi-center Study of the Clinical Outcomes Between Initial CDK 4/6 Inhibitor Plus Endocrine Therapy and Initial Chemotherapy in HR Positive, HER2 Negative Unresectable or Metastatic Breast Cancer in Real World Practice
Brief Title: Initial CDK 4/6 Inhibitor Plus Endocrine Therapy Versus Initial Chemotherapy in HR Positive, HER2 Negative Unresectable or Metastatic Breast Cancer
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Biyun Wang, MD, Professor, Fudan University
Other Study IDs: YOUNGBC-30
Record Dates: First submitted 2024-03-28; First posted 2024-04-03 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer
Keywords: chemotherapy; CDK 4/6 Inhibitor; HR Positive; HER2 Negative
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- CDK 4/6 Inhibitor plus endocrine treatment cohort
- Chemotherapy cohort

SUMMARY:
A multi-center, real world study to evaluate the clinical outcomes between initial CDK 4/6 Inhibitor plus endocrine therapy and initial chemotherapy in HR positive, HER2 negative unresectable or metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. age >= 18 years old;
2. Patients who were diagnosed as HR Positive, HER2 Negative recurrent unresectable (local or regional) or stage IV (M1) breast cancer between June 2020 to October 2023;
3. Received CDK4/6 inhibitor plus endocrine treatment or chemotherapy as first-line therapy for at least one cycle;
4. Complete medical history was available.

Exclusion Criteria:

1. Medical history was incomplete.

Ages: 18 Years to 75 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Patients who were diagnosed as HR Positive, HER2 Negative recurrent unresectable (local or regional) or stage IV (M1) breast cancer between June 2020 to October 2023.
Sampling Method: Non-Probability Sample
Enrollment: 608 (Actual)
Dates: Start 2023-05-20 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
PFS | 6 weeks
  progression-free survival

SECONDARY OUTCOMES:
OS | 6 weeks
  overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Biyun Wang, Professor, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China